CLINICAL TRIAL: NCT05403658
Title: Attrition in Pediatric Obesity Management: A Randomized Feasibility Study
Brief Title: Attrition in Pediatric Obesity Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00111932
Record Dates: First submitted 2022-05-25; First posted 2022-06-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Child Obesity
Keywords: child obesity; clinical care; attrition; childhood obesity; weight management; pediatric; barriers; patient navigation; family navigator
MeSH Terms: conditions — Pediatric Obesity; Tooth Wear

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Study investigators will not know which families were randomized to the experimental group or control group. Data analyses, both quantitative and qualitative, will be led by investigators who will have no direct contact with families and will not have access to information regarding group assignment. Interventions will be delivered by Family Navigators and data collection will be completed by research team members, although both groups will be aware of families' group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Navigation + Usual Care (Experimental): Participants assigned to this arm will receive the Family Navigation (FN) intervention in addition to standard pediatric obesity management (Usual Care).
  Interventions: Behavioral: Family Navigation; Behavioral: Usual Care
- Usual Care (Active Comparator): Participants assigned to this arm will standard pediatric obesity management only.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Family Navigation — FN will be delivered by navigators who will provide support and services that complement obesity management care provided by multidisciplinary teams at the study clinical sites. With advanced training in motivational interviewing and patient- / family-centered care, navigators will access a bundle of logistical and relational strategies to help families derive the greatest possible benefit from their care, which will include working to reduce barriers to care, improve access, and optimize treatment outcomes related to obesity management that is part of their Usual Care. Navigators will provide various resources/supports to study participants including, but not limited to, offering communication via text message, flexible navigator appointments, parking/transit passes, community-based resources, and liaising with members of the multidisciplinary clinical teams at each site.
  Arms: Family Navigation + Usual Care
Behavioral: Usual Care — Usual Care is delivered similarly across the 2 clinical sites. Obesity management is offered by multidisciplinary teams that include clinicians with advanced expertise in pediatrics, nutrition, mental health, physical activity/exercise, and behavior change. Interventions are tailored to families' readiness, capabilities, and motivation to make healthy lifestyle and behavioral changes.

SUMMARY:
Our feasibility study will assess the feasibility and acceptability of Family Navigation (FN) to address attrition (dropout) in pediatric obesity management. Results from this study will help our team to plan a large randomized clinical trial to test the effectiveness of FN in reducing attrition.

The investigators will enroll 108 6-to-17-year-olds enrolled in pediatric obesity management clinics in Calgary, AB and Mississauga, ON (Canada). One-half of the children will receive Family Navigation (FN) + Usual Care (UC) for 12 months; the other half will receive Usual Care only for 12 months. Overall, the study will take 2.5 years to complete.

For children receiving FN, trained navigators will work with children and their families to reduce barriers that limit their access to health services and support. Navigators will offer extra services and resources, such as parking passes for clinic appointments and supportive text messages between appointments. FN is designed to complement the obesity management (Usual Care) received by children and their families. A Steering Committee with children, caregivers, clinicians, and researchers will be created to refine and improve our FN intervention throughout the study.

By having better access to care, children and their families working with navigators may be less likely to drop out and more likely to attend more treatment appointments. Ultimately, the participants may be more likely to achieve success in managing obesity.

DETAILED DESCRIPTION:
Background: Pediatric obesity is prevalent, persistent, and complex. Annual obesity-linked healthcare costs in Canada exceed $7 billion. For people living with obesity, successful obesity management (i.e., reducing or stabilizing weight gain, improving obesity-related consequences) is challenging. Without intervention, obesity and its consequences usually track into adulthood, a pattern that entrenches with increasing obesity severity, underscoring the high value of accessible and effective interventions. Robust evidence demonstrates that multidisciplinary interventions centered on family lifestyle and behavior can help children to manage obesity. However, success is predicted by adhering to treatment regimens, including regularly attending clinical appointments. Effective lifestyle and behavioral interventions require a moderate to high intervention dose (>25 hours of clinic contact over 6-12 months) to optimize benefits (↓BMI, systolic blood pressure; ↑insulin sensitivity, quality of life). Achieving this dose is difficult for families in pediatric obesity management (POM) because many experience barriers and constraints to accessing care, such as schedule availability, transportation costs, and variable motivation. Even the best obesity management interventions are undermined when families discontinue care prematurely. To meet this mandate, the proposed research tackles a common and vexing issue in POM - Attrition.

Purpose: The purpose of this feasibility study is to prepare the study team for a definitive RCT in which the investigators will test the effectiveness of a novel intervention (Family Navigation [FN]) to reduce attrition in 6-17 years old in pediatric obesity management (POM).

Objectives: The primary objectives of the study are to 1) assess children's and caregivers' perceived acceptability of the FN intervention and 2) evaluate attrition and measures of study rigor and conduct, including participant recruitment and enrolment, randomization procedures, and study protocol integrity, against pre-set success indicators. The study's secondary objective is to collect various outcomes (clinical, health services, economics) with established or possible links to attrition for descriptive purposes and hypothesis generation.

Trial Design: The trial is a 2.5-year, multi-method, multi-center randomized feasibility study that has 2 arms and follows parallel assignment. Children will be assigned to an experimental or control group after they enroll in multidisciplinary POM clinics in Calgary, AB and Mississauga, ON (Canada).

Trial Interventions: The experimental group will receive FN + Usual Care. FN will be co-designed to reduce attrition by managing barriers and eliminating constraints that limit access to care. FN increases access to a moderate to high intervention dose, increasing success in POM. The control group will receive Usual Care only (delivered similarly in the 2 study clinics).

Co-designing Family Navigation, a child- and family-centered intervention: Over the past decade, the investigators collected and synthesized qualitative and quantitative data on attrition from hundreds of families and clinicians. Equipped with this knowledge and experience, the investigators now apply it, working in partnership with the study Steering Committee (SC) to continue co-designing the FN intervention. The trial's participatory approach draws on key elements of Experience-Based Co-Design, an orientation that focuses on understanding SC members' experiences with health services, identifying potential improvements, and making changes together. With co-design, the investigators plan to increase intervention relevance and appropriateness, bringing together people who possess experiential knowledge (children, caregivers) with people who have expert knowledge (clinicians, researchers); the 2 knowledge systems enrich each other. The investigators have substantial experience in co-designing and refining health services and interventions in partnership with stakeholders; the current study extends the research team's legacy of collaborative, engaged research.

SC organization: The SC structure and values align with expert recommendations for stakeholder-engaged research. From the 2 POM clinics, the investigators will recruit 3 13-to 17-year-olds and 3 caregivers with first-hand experience in managing obesity, 3 clinicians working in POM, and one clinic manager, all of whom will join the research team members on the committee.

Delivering FN: The SC will optimize FN delivery, determining the most practical and important elements, a critical task for future scalability and sustainability. Each of the 2 study clinics will have a navigator to deliver FN. Navigators will be trained and equipped with resources for individualized support to benefit families in POM. Navigators will start by orienting families to the intervention and completing a detailed needs assessment, highlighting areas for support to manage barriers and remove constraints to POM access. Navigators will access a bundle of logistical and relational strategies to help families remove constraints or manage barriers in access to POM care. These multiple evidence-based strategies emerged from the investigators' attrition research with families and clinicians, but none are provided currently in our 2 clinics.

Logistical Strategies in FN:

* Communication via text message. Navigators will connect with families by study-dedicated smartphones to schedule appointments (book, remind, coordinate care), celebrate successes, troubleshoot barriers and constraints to care and share educational resources.
* Flexible navigator appointments. Beyond their POM visits, families and navigators will meet at convenient times, including evenings and weekends. Most appointments will be virtual (videoconference, phone), with in-person visits returning during the study term, pandemic permitting.
* Parking/Transit passes (up to 16 for in-person clinic visits). Passes will be used for any in-person visits of families with navigators and POM clinicians (or researchers).
* Community-based resources. Navigators will build a list of resources and services (e.g., mental health support, school-based programs) for families in Calgary and Mississauga.

Relational Strategies in FN: Navigators will use motivational interviewing (MI) principles, a directive, client-centered counseling approach used in most navigation interventions. Navigators will focus on listening to and validating family challenges, exploring the desire to continue POM. In some cases, they will work intensively with families, liaising regularly with clinicians to integrate care. In other cases, they will interact with families exclusively. Family preferences and needs drive appointment frequency with navigators: weekly, biweekly, or monthly; virtual (videoconference or phone) or in-person, pandemic permitting; 30-60 min long. As a tailored intervention, FN acknowledges that the desire to maximize POM adherence varies by family and that ambivalence is common in managing obesity. Navigator-family discussions may include children and caregivers together or separately, based on preferences and needs. Navigators will adhere to a communication and documentation protocol if families disclose information (e.g., child safety) beyond their scope.

Usual Care: The control intervention is Usual Care for POM, delivered similarly across our 2 clinics by multidisciplinary teams who follow family-centered care principles and guidelines. At clinic presentation, children will complete a comprehensive health assessment to inform lifestyle (diet, physical activity, sedentary habits, sleep) and behavioral goal setting and subspecialty medical referrals, if indicated. Children and caregivers attend POM visits regularly to make and maintain healthy changes. Appointments with physicians occur at least every 6 months and more frequently with other clinicians (e.g., RD, Psych). The dose and duration of POM vary according to family need, motivation, and illness severity. The 2 study clinics offer 1-on-1 virtual care by videoconference or phone, with in-person visits restarting, pandemic permitting. Families attend most visits in their first 3-6 months, with appointment frequency decreasing over time, consistent with guidelines.

Sample Size: The investigators will recruit 108 participants (54/group; 54/site). Feasibility studies do not include formal sample size calculations, but experts recommend 12-36/arm. So, the investigators will enroll 27/arm/site.

Recruitment: Research assistants will work with clinical teams to give families details about the study at clinic enrolment. The research team expects families to have an interest in this study because they have the potential to benefit directly from study participation via FN. Recruitment will span ~12 months.

Number of Centers: The study has 2 multidisciplinary, Canadian POM clinic sites: Calgary, AB (Alberta Children's Hospital) and Mississauga, ON (Trillium Health Partners).

ELIGIBILITY:
Inclusion Criteria:

* be 6-17 years old,
* have a BMI ≥97th percentile,
* have a primary caregiver (parent/guardian) agree to participate

Exclusion Criteria:

* participants will be excluded if caregivers cannot communicate in English since the Family Navigation intervention will be available in English only.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Perceived acceptability of Family Navigation (Child) | 3, 6, and 12 months post-baseline
  The investigators will complete semi-structured, 1-on-1 interviews with children using appropriate interview guides. Guides are based on multiple domains of intervention acceptability according to the Theoretical Framework of Acceptability, which includes multiple component constructs. Our sampling uses age as a proxy for developmental stage (6-9y; 10-13y; 14-17y). Groupings were based on developmental differences that could influence participants' perceptions and experiences of the Family Navigation intervention. Children from (10-13y) and (14-17y) age groups will be interviewed. For the 6-9y group, no children will be interviewed; however, their caregivers will be interviewed. Interviews will be recorded, undergo voice-to-text conversion, or be transcribed verbatim. Perceived acceptability among children will be measured in a sub-set of the families in the FN + UC group.
Perceived acceptability of Family Navigation (Caregiver) | 3, 6, and 12 months post-baseline
  The investigators will complete semi-structured, 1-on-1 interviews with caregivers, using interview guides that are appropriate for them. Guides are based on multiple domains of intervention acceptability according to the Theoretical Framework of Acceptability, which includes multiple component constructs. Sampling for caregivers' interviews will be performed considering their children's age group. Our sampling uses the age of the children as a proxy for developmental stage (6-9y; 10-13y; 14-17y). Groupings were based on developmental differences that could influence participants' perceptions and experiences of the Family Navigation intervention. Interviews will be recorded, undergo voice-to-text conversion, or be transcribed verbatim. Perceived acceptability among children will be measured in a sub-set of the families in the FN + UC group.

SECONDARY OUTCOMES:
Sociodemographic data | Baseline
  The investigators will collect the following sociodemographic data using a standardized case report form: Dates of birth (child and caregiver), the relationship between child and caregiver, ethnicity (child and caregiver), and socioeconomic status (by caregiver self-report).
Measures of study rigor and conduct | Baseline
  The investigators will use a standard approach to document eligible, approached, recruited, and enrolled participants to generate counts and rates and work with clinic staff on procedures to maximize study awareness for all families. The thresholds for pre-set success indicators were decided based on objective criteria (when possible) and experience gained through study implementation as well as data analysis and interpretation with Stakeholder Committee and research team.
Attrition | 3, 6, and 12 months post-baseline
  The operational definition of attrition in the study includes 'yes'/'no'/'unknown' categories. If a child discontinues pediatric obesity management at any point up to 12 months post-baseline or if an appointment is missed or canceled without rescheduling and the investigators have no follow-up communication with the family after 4 phone/text messages over 4 weeks and no scheduled upcoming appointments, they will be classified as 'yes'. If a child remains in pediatric obesity management at 12 months post-baseline, they will be classified as 'no'. If a child's status cannot be confirmed, they will be classified as 'unknown'. The pre-set success indicators or threshold for attrition is 15%-25% for the experimental group (FN+ UC) and 30%-40% for the control group (UC only). These thresholds are decided based on objective criteria (when possible) and experience gained through study implementation as well as data analysis and interpretation with Stakeholder Committee and research team.
PedsQL | Baseline, 3, 6, and 12 months post-baseline
  Health-related quality of life questionnaire - assessed by children (self-report) and caregivers (proxy report)
Child- and caregiver-reported internalized and experienced weight bias | Baseline, 3, 6, and 12 months post-baseline
  Survey to assess child- and caregiver-reported internalized and experienced weight bias
Working Alliance Inventory | Baseline, 3, 6, and 12 months post-baseline
  Survey to quantify the strength of therapy relationship between caregivers and navigators/clinicians
Family treatment expectations for obesity management | Baseline
  Survey to assess family treatment expectations for obesity management
Child and caregiver motivation to change lifestyle habits | Baseline, 3, 6, and 12 months post-baseline
  Survey to assess child and caregiver motivation to change lifestyle habits
PedsQL Healthcare Satisfaction | Baseline, 3, 6, and 12 months post-baseline
  Questionnaire to assess caregiver-rated quality of care.
Unintended consequences of treatment | Baseline, 3, 6, and 12 months post-baseline
  Survey to assess unintended consequences of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Ball, PhD RD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ball GDC, O'Neill MG, Noor R, Alberga A, Azar R, Buchholz A, Enright M, Geller J, Ho J, Holt NL, Lebel T, Rosychuk RJ, Tarride JE, Zenlea I. A multi-center, randomized, 12-month, parallel-group, feasibility study to assess the acceptability and preliminary impact of family navigation plus usual care versus usual care on attrition in managing pediatric obesity: a study protocol. Pilot Feasibility Stud. 2023 Jan 23;9(1):14. doi: 10.1186/s40814-023-01246-w. PMID 36691103